CLINICAL TRIAL: NCT06374381
Title: Adaptive Trial of Parent Empowerment and Coaching in Early Intervention: PEACE for ImPACT Study
Brief Title: PEACE for ImPACT Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency); Michigan State University (Other)
Responsible Party: Principal Investigator, Melanie Pellecchia, PhD, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 854990
Record Dates: First submitted 2024-03-19; First posted 2024-04-18 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Early Intervention; Caregiver Mediated Interventions; Caregiver or Parent Coaching
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to randomization condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adherent: Continue Online Resources (No Intervention): Providers who are adherent to parent coaching strategies during the 8 and 16 week timepoints will not be randomized and continue to use the PEACE Online Resources. They will not receive further implementation supports.
- Non Adherent: Continue Online Resources (Placebo Comparator): After 8 and 16 weeks, providers with low coaching adherence could be randomized to continue using the PEACE online resources with no further implementation supports.
  Interventions: Behavioral: PEACE Online Resources
- Non Adherent: Group Facilitation (Experimental): After 8 and 16 weeks, providers with low coaching adherence could be randomized to receive weekly group facilitation.
  Interventions: Behavioral: PEACE Weekly Group Facilitation
- Non Adherent: Individual Facilitation (Experimental): After 16 weeks, providers may be randomized to receive individual facilitation with an expert coach if they continue to be non adherent to the use of parent coaching strategies.
  Interventions: Behavioral: PEACE Weekly Individual Facilitation

INTERVENTIONS:
Behavioral: PEACE Online Resources — The PEACE online resource includes self-paced training modules that cover the foundations of caregiver coaching, caregiver perspectives towards coaching, strategies for aligning with caregivers and gaining buy-in for coaching, evidence-based strategies to empower caregivers from marginalized backgrounds, and strategies to improve collaboration and cohesion among providers working with the same child. Each module includes brief example videos, easy-to read infographics, tip sheets, and checklists to guide implementation. A virtual communication application, Slack, facilitates frequent communication, enhances social networks among providers, and creates social norms related to the use of caregiver coaching. Providers can post questions or suggestions, share resources, and receive updates about other providers' accomplishments. Consultants frequently post encouraging messages and progress updates to increase motivation and shared norms for coaching.
  Arms: Non Adherent: Continue Online Resources
Behavioral: PEACE Weekly Group Facilitation — Facilitation comprises interactive problem solving and support, a shared understanding of need for improvement, and a supportive interpersonal relationship. Providers participate in 12 weekly group facilitation meetings for one hour virtually with an expert consultant focused on auditing providers' fidelity to caregiver coaching through role-play and performance feedback. Each group meeting aligns with content from the PEACE online resource library modules.
  Arms: Non Adherent: Group Facilitation
Behavioral: PEACE Weekly Individual Facilitation — Individual facilitation is delivered virtually for one hour each week for eight weeks with a consultant focused on reflection and problem solving any identified implementation barriers, as well as practice and performance feedback.
  Arms: Non Adherent: Individual Facilitation

SUMMARY:
Investigators will test the impact of the PEACE implementation toolkit and determine the level of implementation support needed to improve early intervention providers use of caregiver coaching with families of young children with autism who receive early intervention services. The study will also assess caregiver and child outcomes for families receiving caregiver coaching and the cost effectiveness of the PEACE implementation toolkit. The investigators will enroll 200 early intervention providers, and 400 parent-child dyads.

DETAILED DESCRIPTION:
Investigators are partnering with the two early intervention systems and their respective agencies in Philadelphia that serve young children receiving early intervention services under the age of 5. Investigators will enroll 200 early intervention providers who deliver services to young children in Philadelphia. All providers will receive training on Project ImPACT. The investigators will also recruit 400 parent-child dyads from participating providers' caseloads and follow them over a 6 month period. Providers will be given access to the PEACE Implementation Toolkit to aid their implementation of Project ImPACT with enrolled families. At week 8, providers caregiver coaching fidelity with enrolled families will be assessed. Non-adherent providers will be randomized to either 1) continue using the PEACE Online Resources or 2) receive added support through 8 weeks of group facilitation with an EI consultant. The fidelity assessment will occur again at week 16 of the intervention. Non-adherent providers will be re-randomized to either 1) continue using the PEACE Online Resources, 2) receive 8 weeks of group facilitation with an EI consultant or 3) receive 8 weeks of individual facilitation with an EI consultant. At week 24 investigators will assess implementation fidelity for a final time. Secondary outcomes related to caregiver and child outcomes will be assessed at baseline and week 24. Planned analyses for all research questions can be found in the research study protocol available for review.

Completion of this project could radically transform the Philadelphia EI system's capacity to implement caregiver coaching with families of young children with ASD by providing critical supports to historically marginalized families, thereby improving learning trajectories for many young children with ASD. Data gathered through this project will be directly generalizable to EI systems across the country and inform the large-scale implementation of caregiver-mediated interventions for ASD within other publicly funded EI systems.

ELIGIBILITY:
Inclusion Criteria:

1. Provider is employed by a Philadelphia EI agency
2. Provider has > 5 children with/at risk for ASD on their caseload.
3. Child is receiving EI services from a participating provider.
4. Child has a classification of ASD or high ASD risk as determined by the EI system.
5. Child is not transitioning from EI services for at least 6 months.
6. Caregiver speaks English or Spanish (Project ImPACT materials are available in Spanish).
7. Caregiver is willing to participate in weekly coaching sessions.

Exclusion Criteria:

1. Participants will be excluded if they do not speak English or Spanish, as the published intervention materials are currently available in English and Spanish and the research team is able to communicate with participants in English or Spanish only.

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Parent Empowerment and Coaching in Early Intervention (PEACE) Caregiver Coaching Fidelity Tool | Weeks 8, 16, and 24 weeks of intervention
  The tool consists of 25 items, rated on a 5-point scale with a rating of 4 or 5 indicating acceptable adherence. A score of 80% indicates adherence on the overall measure (i.e., 80% of the items rated at 4 or 5).

SECONDARY OUTCOMES:
Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO) | 6 months (Baseline and Week 24)
  The PICCOLO is a checklist of 29 observable, developmentally supportive parenting behaviors with children ages 10-47 months. The PICCOLO has four domains: Affection, Responsiveness, Encouragement, and Teaching. Total scores on each domain are used to monitor change in parenting behaviors. The minimum score is a 0 and a maximum score is 58. Higher scores indicate higher occurrences of supportive behaviors.
Autism Impact Measure (AIM) | 6 months (Baseline and Week 24)
  A 41-item parent report questionnaire designed to track incremental change in frequency and impact of core ASD symptoms. The frequency and impact of symptoms are determined by a 5-point scale. Higher scores on the measure indicate greater symptom severity.
Social Communication Checklist (SCC) | 6 months (Baseline and Week 24)
  A 47-item parent report checklist that is used as part of the Project ImPACT program to help parents set their child's social communication goals and assess child progress. An initial psychometric evaluation suggests that it is reliable, sensitive to change after intervention, and strongly related to well-established measures of social-communication functioning. Respondents indicate whether a child uses a specific skill on a 3-point scale. Scores are summed for domain scores (Social Engagement, Expressive Communication, Receptive Communication, and Imitation/Play) and a Total Score. Higher scores indicate that skills are being used more frequently.
Confusion, Hubbub, and Order Scale (CHAOS) | Baseline
  A validated parent-report measure of disorder and chaos in the home will be used to measure home environmental factors that may interfere with the use of caregiver coaching. Responses are formatted as a True/False or Yes/No format. Once completed, the 15 items are summed for a Total Score. A higher score indicates more chaotic, disorganized, and hurried characteristics of the home.
Acceptability, Appropriateness, and Adoption measure | 6 months (Week 24)
  A measure that specifically queries for respondents views about the usefulness, acceptability, and the extent to which they used the components of the toolkit. Respondents rate the toolkit's acceptability, appropriateness, and their use of the components on a 5-point scale. Higher scores indicate higher levels of acceptability, appropriateness, and adoption.
Qualitative Interview | 6 months (Week 24)
  We will conduct qualitative interviews with 20% of the early intervention providers in each cohort. We will interview them using an interview guide with questions eliciting feedback on the PEACE Implementation Toolkit and the implementation supports that were provided.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Pellecchia, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Mental Health, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT06374381/Prot_SAP_000.pdf